CLINICAL TRIAL: NCT00689650
Title: Fractional Nonablative 1540 nm Laser Resurfacing for Burn Scars- A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Other Study IDs: H-D-2007-0094
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Burn Scar Patients

ARMS (2):
- A (Experimental)
  Interventions: Device: 1540 nm fractional laser
- B (No Intervention)

INTERVENTIONS:
Device: 1540 nm fractional laser
  Arms: A

SUMMARY:
The objective was to evaluate the efficacy of 1540 nm fractional laser treatment of mature burn scars.

ELIGIBILITY:
Inclusion Criteria:

* Burn scars with and without previous skin grafting.

Exclusion Criteria:

* A tendency to produce hypertrophic scars or keloids,
* Previous treatment with dermabrasio, chemical peel, filler, laser treatment or Intense Pulsed Light (IPL) of study areas,
* Photosensitivity,
* Pregnancy or lactation,
* Current anticoagulative medication,
* Oral retinoid drugs within the past 6 months,
* Pigmentation after recent exposure to sun or solarium,
* Patients not considered to be able to follow the treatment protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-11

PRIMARY OUTCOMES:
Change of skin texture from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg University Hospital, Copenhagen NV, Denmark